CLINICAL TRIAL: NCT02101190
Title: Open-label, Single-dose, Multi-center Study, Investigating the Pharmacokinetics of BIA 9-1067 in Subjects With Hepatic Impairment
Brief Title: Pharmacokinetics of BIA 9-1067 in Subjects With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIA-91067-106
Record Dates: First submitted 2012-01-20; First posted 2014-04-02 (Estimated); Results first posted 2015-01-15 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Parkinson's Disease
Keywords: BIA 9-1067; Opicapone; catechol-O-methyltransferase (COMT)
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 - Hepatic impaired subjects (Experimental): Group 1 - subjects with moderate chronic hepatic impairment treated with BIA 9-1067
  Interventions: Drug: BIA 9-1067
- Group 2 - Healthy subjects (Experimental): Group 2 - healthy subjects treated with BIA 9-1067
  Interventions: Drug: BIA 9-1067

INTERVENTIONS:
Drug: BIA 9-1067 — Opicapone, OPC
  Other Names: Opicapone

SUMMARY:
The purpose of this study is to assess the pharmacokinetics (PK) of BIA 9-1067 in patients with moderate chronic hepatic impairment and in matched healthy subjects.

DETAILED DESCRIPTION:
This was an open-label, single-dose, parallel-group, in-patient, nonrandomized study conducted in 8 patients with moderate chronic hepatic impairment and in 8 healthy matched subjects matched by origin, age, sex, weight, and smoking habits.

Each hepatic impaired patient and matched healthy subject participated in the study for approximately one month, including a 21-day screening period and a 4-day/4-night inpatient period. The inpatient period covered the period from Day -1 to Day 4 morning (through 72 hours after administration). The final study evaluation was performed for all subjects in the morning of the day of discharge, Day 4.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

1. Men or non-lactating and non-pregnant women,
2. Women of non-childbearing potential (WONCBP), expected to be surgically sterile (hysterectomy, oophorectomy, or tubal ligation) or postmenopausal for >1 year,
3. Women of childbearing potential (WOCBP), expected to be using an acceptable method of contraception (sexual abstinence, implants, IUD, injectables, vasectomised partner or association of condom + spermicide, diaphragm + spermicide, diaphragm + condom) for a period of at least 1 month before and after dose administration. WOCBP were expected to have a negative pregnancy test (serum beta-human chorionic gonadotropin [β-HCG]) result within 48 hours before the start of the first IMP administration. Hormonal contraceptives were not allowed because the effect of BIA 9-1067 on the metabolism of oral contraceptives and vice versa is not yet known,
4. Male subjects should not have been planning to father a child or donate sperm, during the study and 1 month after the end of the study. Acceptable methods of contraception comprised condom and a medically accepted contraceptive method for the female partner (intra-uterine device with spermicide, hormonal contraceptive for the last 2 months),
5. Expected to have a high probability for compliance with and completion of the study, Hepatic Impaired Patients only:
6. Aged 18 to 65 years,
7. Body weight ≥ 50 kg,
8. Child Pugh class B (score at 7, 8 or 9) calculated according to the Child-Pugh classification based on history, physical examination, and laboratory test results at screening and on Day -1,
9. Hepatic impairment should not have been associated to an underlying systemic disease,
10. Medications necessary for the management of the hepatic disease or concomitant conditions were permitted if the therapeutic regimen has been stable for at least 7 days before BIA 9-1067 administration and if they did not interfere with the kinetics of the tested product,

    Matched Healthy Subjects only:
11. Aged 18 to 65 years,
12. Body weight ≥ 50 kg,
13. Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and 12-lead electrocardiogram (ECG). Alanine aminotransferase (ALT) and creatinine levels should have been strictly within the normal range for eligibility.

Exclusion Criteria:

1. Presence or history of any disorder that may prevent the successful completion of the study. Allergies and Adverse Drug Reactions
2. History of multiple and/or severe allergies to drugs or foods or a history of anaphylactic reactions.
3. Known or suspected allergy or other adverse drug reactions to the trial product or related products (e.g tolcapone or entacapone).
4. Positive pregnancy test result (serum Beta-HCG) for women of childbearing potential only.
5. Consumption of any caffeine-containing products (eg, coffee, tea, chocolate, or cola), grapefruit, grapefruit-containing products, or alcoholic beverages from 48 hours before study day 1 until the end of the inpatient confinement period.
6. Involvement in other investigational studies of any type within 30 days of BIA 9-1067 administration.
7. Donation of blood within 90 days of study day 1.
8. Evidence of unstable clinically significant disease other than impaired hepatic function (e.g., cardiovascular, cerebrovascular, respiratory, renal disease, or any serious disorder that currently requires a physician's care).
9. Recent history or presence of any disorder that may interfere with the absorption, distribution, metabolism, or excretion of BIA 9-1067 (except hepatic impairment).
10. Patients with severe encephalopathy.
11. Acute exacerbation of hepatic disease, as indicated by worsening of clinical and/or laboratory signs of hepatic impairment, within the 2 weeks before BIA 9-1067 administration (eg, advanced ascites, infection of ascites, fever, hepatic encephalopathy or active gastrointestinal bleeding (hematemesis, melena), significant abdominal pain, persistent nausea and vomiting, or a worsening of total bilirubin or prothrombin time by >50%).
12. Presence of a hepatocellular carcinoma, or an acute hepatic disease caused by infection or drug toxicity.
13. Presence of surgically created portal-systemic shunt.
14. Positive serologic finding for human immunodeficiency virus (HIV) antibodies.
15. Prescription and over-the-counter (OTC) medication doses must be stable for 7 days before IMP administration.

    Healthy Matched Subjects only:
16. History of alcoholism or excessive daily alcohol consumption within the past year. Excessive alcohol consumption is regarded as an average weekly intake of more than 14 units for women and 21 units for men (1 unit of alcohol = 8 to 10 g and is approximately equivalent to 1 glass of wine or 250 mL of beer or a standard measure of spirits).
17. Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
18. Any clinically important deviation from normal limits in physical examination, vital signs, or 12-lead ECGs.
19. Acute disease state (e.g., nausea, vomiting, fever, diarrhea) within 7 days of study day 1.
20. Positive serologic findings for HIV antibodies, hepatitis B surface antigen (Hbs Ag), and/or hepatitis C virus (HCV) antibodies.
21. Recent history or presence of any disorder that may interfere with the absorption, distribution, metabolism, or excretion of BIA 9-1067.
22. Use of any prescription drug within 30 days of IMP administration.
23. Use of any OTC drugs including herbal supplements (except for the occasional use of acetaminophen and vitamins ≤100% recommended daily allowance) within 14 days of study day 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricio Soares-da-Silva, MD, PhD, Study Director — BIAL - Portela & Cª, S.A.
Locations (3):
- Biotrial, 7-9 rue Jean-Louis Bertrand, Rennes, France
- Russia (2):
  - City clinical Hospital N°64, Moscow, Moscow
  - City clinical Hospital N°3, Moscow, Moscow

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 - Hepatic Impaired Subjects | Group 2 - Healthy Subjects
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - Hepatic Impaired Subjects | Group 2 - Healthy Subjects | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Plasma Concentration of BIA 9-1067
Description: BIA 9-1067 Cmax following a single dose of 50mg BIA 9-1067
Time Frame: pre-dose (within 1 hour before dose administration) and then at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 60 and 72 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1 - Hepatic Impaired Subjects | Group 2 - Healthy Subjects
Number analyzed (Participants) | 8 | 8
ng/mL | 1108 (448) | 559 (119)

2. Primary Outcome: Tmax - Time to Reach Cmax
Description: BIA 9-1067 Tmax following a single dose of 50mg BIA 9-1067
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Group 1 - Hepatic Impaired Subjects | Group 2 - Healthy Subjects
Number analyzed (Participants) | 8 | 8
hours | 3.0 [1.5 to 4.0] | 3.0 [1.5 to 4.0]

3. Primary Outcome: Area Under the Curve (AUC0-t)
Description: BIA 9-1067 AUC0-t following a single dose of 50mg BIA 9-1067
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng.hr/mL
Arm/Group | Group 1 - Hepatic Impaired Subjects | Group 2 - Healthy Subjects
Number analyzed (Participants) | 8 | 8
ng.hr/mL | 3392 (1584) | 1724 (503)

ADVERSE EVENTS:
Arm/Group | Group 1 - Hepatic Impaired Subjects | Group 2 - Healthy Subjects
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 - Hepatic Impaired Subjects (N=8) | Group 2 - Healthy Subjects (N=8)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other